CLINICAL TRIAL: NCT04281316
Title: Impact of Nasal High Flow (NHF) Versus Home Non-invasive Ventilation (NIV) on Nocturnal Transcutaneous PCO2 (PtCO2) in Stable COPD Patients: A Non-inferiority Study
Brief Title: High-Flow in Hypercapnic Stable COPD Patients
Acronym: HIGH-FLOW
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack enrollment
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Icadom (Industry); Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38R19.250
Record Dates: First submitted 2020-02-11; First posted 2020-02-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Adherence, Treatment
Keywords: non-compliance; NIV; NHF; COPD; hypercapnic respiratory failure
MeSH Terms: conditions — Treatment Adherence and Compliance; Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Invasive Ventilation device group (Active Comparator): The patients in the NIV arm will receive treatment as in their usual care with an additional educational session of one hour for improving compliance.
  Interventions: Device: Non Invasive Ventilation; Other: Education session
- Nasal High Flow (MyAirvo) device group (Experimental): The patients in the NHF arm will receive NHF treatment and two hours training adaptation session will be conducted in the hospital.
  Interventions: Device: Nasal High Flow installation; Other: Training session

INTERVENTIONS:
Device: Nasal High Flow installation — Participants randomized in NHF group will receive the nasal high flow (NHF) treatment delivered by myAirvo2.
  Nasal High-Flow (NHF) is a treatment delivering heated, humidified, and optionally oxygen-enriched, air at high flow rates through a nasal cannula. The physiologic effects of NHF are an improvement in gas exchanges including a reduction in hypercarbia an optimization in breathing patterns with a reduction of work of breathing and high compliance as delivered via a comfortable nasal interface
  Other Names: MyAirvo Device
  Arms: Nasal High Flow (MyAirvo) device group
Device: Non Invasive Ventilation — Participants randomized in the Non Invasive Ventilation group will receive treatment as in their usual care.
  Arms: Non Invasive Ventilation device group
Other: Training session — The patients in the Nasal High Flow (MyAirvo) arm will receive two hours training adaptation session in the hospital
  Arms: Nasal High Flow (MyAirvo) device group
Other: Education session — Participants randomized in the Non Invasive Ventilation group will receive an additional educational session of one hour for improving compliance.
  Arms: Non Invasive Ventilation device group

SUMMARY:
Monocentric, prospective, open, randomized 1:1, controlled study to evaluate the impact of nasal high-flow (NHF) on nocturnal transcutaneous PCO2 (PtCO2) compared to non-invasive ventilation ± Long-Term Oxygen Therapy (LTOT) in patients with a Chronic obstructive pulmonary disease (COPD)-related hypercapnic respiratory failure.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a growing global health concern, causing considerable health-related costs and increased mortality. COPD is nowadays considered a complex, heterogeneous and systemic condition.

In the late stage of the disease, non-invasive ventilation (NIV) is widely prescribed either to treat acute hypercapnic respiratory failure during COPD exacerbations or for long term home management.

A meta-analysis has shown that higher daytime PaCO2 occurred in home NIV treated COPD patients when NIV compliance is less than 5 h/day. Thus, an optimal NIV adherence is a key target for controlling nocturnal and diurnal hypoventilation and improving prognosis.

COPD is the clinical scenario during which a good NIV adherence is difficult to achieve. Particularly, in COPDs exhibiting hyperinflation, NIV can aggravate dynamic hyperinflation resulting in unrewarded inspiratory efforts, poor sleep and low NIV compliance. Alternatives to NIV are then desirable in this specific subgroup of hypercapnic COPD with poor adherence to NIV.

During this trial, stable COPD patients treated by long term home Non-Invasive Ventilation (NIV) treatment following French national recommendations and exhibiting a NIV compliance of (less than 5 hours and more than 1 hour) per day in the last 3 months prior to inclusion will be randomized via a secure electronic website to either continue with their current NIV treatment or receive the nasal high flow (NHF) treatment delivered by myAirvo2 during 3 months Nasal High-Flow (NHF) is a treatment delivering heated, humidified, and optionally oxygen-enriched air at high flow rates through a nasal cannula. The main physiologic effects of NHF are an improvement in gas exchanges including a reduction in hypercapnia, an optimization in breathing patterns with a reduction of work of breathing. Nasal High-Flow (NHF) is delivered via a comfortable nasal interface and has demonstrated good treatment adherence.

The investigators hypothesize that in COPD-related hypercapnic chronic respiratory failure with limited compliance to NIV (less than 5 hours per night), nasal High-Flow (NHF) will be non-inferior for controlling nocturnal hypoventilation and might improve daytime subjective patients centered outcomes, physical activity and nocturnal adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD (FEV1/FVC < 70%) and long term indication for home NIV for initiated at least 3 months prior the inclusion.
* Compliance with NIV (less than 5 hours and more than 1 hour) per night on average during the last 3 months prior to inclusion.
* Naïve to Nasal High Flow (NHF) therapy, i.e. having not used NHF in the last 6 months prior to inclusion.
* Able to understand, follow objectives and methods of protocol in French language.
* Patient affiliated to social security insurance or beneficiary of social health insurance.
* Willing and able to give written Informed Consent and to comply with the requirements of the study protocol.

Exclusion Criteria:

* Significant uncontrolled cardiac disease (investigator judgment), and/or Left Ventricular Ejection Fraction (LVEF) < 45%.
* Known co-existing obstructive sleep apnea requiring expiratory pressure above 6 cmH20.
* Severe nasal obstruction, previous upper airway surgery preventing the usage of NHF, or, at the discretion of investigator, any other contraindication for using the NHF.
* Patients who are unable or unwilling to give informed consent.
* Participating in another research study.
* Patient protected by the Law, under guardianship or curators.
* Pregnancy and nursing mothers
* Patient not covered by a health insurance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Changes on nocturnal parameters with the nasal high-flow (NHF) compared to non-invasive ventilation in patients with a COPD-related hypercapnic respiratory failure. | between night at day 1 (baseline) and night at day 90 (3 months after)
  Differences in mean overnight transcutaneous PtCO2 measurement

SECONDARY OUTCOMES:
Evaluation the impact of nasal high-flow (NHF) on other nocturnal parameters compared to non-invasive ventilation ± LTOT compared to non-invasive ventilation in patients with a COPD-related hypercapnic respiratory failure. | between night at day 1 (baseline) and night at day 90 (3 months after)
  Maximum PtCO2
Treatment adherence | between night at day 1 (baseline) and night at day 90 (3 months after)
  Treatment adherence measured objectively by download of NIV software data and for NHF (myAirvo2) by hour meter & daily average of usage (screen display)
Daytime blood gas values in ambient air | between day 0 (inclusion) and day 97 (end of the study)
  PaCO2 & PaO2 in ambient air will be measured by blood gas sample in NHF group compared de NIV group
Other nocturnal parameter | between night at day 1 (baseline) and night at day 90 (3 months after)
  Overnight Sp02 will be evaluated by nocturnal oximetry at home in order to determine: mean nocturnal SaO2, nadir nocturnal SaO2, cumulative time spent below 90% of SaO2 (CT<90%), Oxygen Desaturation Index.
Physical activity | for 7 days from the day 1 and for 7 days from the day 90
  An actimetry will allow evaluating physical activity (number of steps)
Sleep activity | between night at day 1 (baseline) and night at day 90 (3 months after)
  An actimetry will allow evaluating total sleep time in minutes
Sleep activity | between night at day 1 (baseline) and night at day 90 (3 months after)
  An actimetry will allow evaluating sleep onset latency in minutes
Sleep activity | between night at day 1 (baseline) and night at day 90 (3 months after)
  An actimetry will allow evaluating sleep efficiency
Pulmonary function tests | between day 0 and day 97
  Pulmonary function will be evaluated by routine patient care spirometry and will measure Vital capacity (VC) in liters
Pulmonary function tests | between day 0 and day 97
  Pulmonary function will be evaluated by routine patient care spirometry and will measure Forced vital capacity (FVC) in liters
Pulmonary function tests | between day 0 and day 97
  Pulmonary function will be evaluated by routine patient care spirometry and will measure Forced expiratory volume (FEV) in liters
Health related quality of life | between day 0 and day 97
  Subjective functioning and quality of life will be measured by self-reporting questionnaire EQ-5D-5L
Health related quality of life | between day 0 and day 97
  Subjective functioning and quality of life will be measured by self-reporting questionnaire SGRQ
Cardiovasculary function | between day 0 and day 97
  Blood pressure measurements will be done three times during rest at five minutes intervals to provide informations on systolic, diastolic and mean blood pressure
Number of participants with adverse events will be assessed in each group by interrogating patients in order to assess the safety of nasal high-flow (NHF) treatment | between day 0 and day 97
  All safety data will be recorded through an Electronic Medical Record as reported by the patient or recorded by the research nurse

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, MD PhD, Principal Investigator — Laboratoire EFCR, CHU de Grenoble
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biener AI, Decker SL, Rohde F. Prevalence and Treatment of Chronic Obstructive Pulmonary Disease (COPD) in the United States. JAMA. 2019 Aug 20;322(7):602. doi: 10.1001/jama.2019.10241. No abstract available. PMID 31429884
- [Background] Riley CM, Sciurba FC. Diagnosis and Outpatient Management of Chronic Obstructive Pulmonary Disease: A Review. JAMA. 2019 Feb 26;321(8):786-797. doi: 10.1001/jama.2019.0131. PMID 30806700
- [Background] Houben-Wilke S, Augustin IM, Vercoulen JH, van Ranst D, Bij de Vaate E, Wempe JB, Spruit MA, Wouters EFM, Franssen FME. COPD stands for complex obstructive pulmonary disease. Eur Respir Rev. 2018 Jun 6;27(148):180027. doi: 10.1183/16000617.0027-2018. Print 2018 Jun 30. PMID 29875138
- [Background] Suh ES, Murphy PB, Hart N. Home mechanical ventilation for chronic obstructive pulmonary disease: What next after the HOT-HMV trial? Respirology. 2019 Aug;24(8):732-739. doi: 10.1111/resp.13484. Epub 2019 Feb 7. PMID 30729638
- [Background] Crimi C, Noto A, Princi P, Cuvelier A, Masa JF, Simonds A, Elliott MW, Wijkstra P, Windisch W, Nava S. Domiciliary Non-invasive Ventilation in COPD: An International Survey of Indications and Practices. COPD. 2016 Aug;13(4):483-90. doi: 10.3109/15412555.2015.1108960. Epub 2016 Jan 8. PMID 26744042
- [Background] Kohnlein T, Windisch W, Wegscheider K, Welte T. Non-invasive positive pressure ventilation for severe COPD--Authors' reply. Lancet Respir Med. 2014 Oct;2(10):e19. doi: 10.1016/S2213-2600(14)70215-2. No abstract available. PMID 25298063
- [Background] Murphy AM, Thomas A, Crinion SJ, Kent BD, Tambuwala MM, Fabre A, Pepin JL, Roche HM, Arnaud C, Ryan S. Intermittent hypoxia in obstructive sleep apnoea mediates insulin resistance through adipose tissue inflammation. Eur Respir J. 2017 Apr 19;49(4):1601731. doi: 10.1183/13993003.01731-2016. Print 2017 Apr. PMID 28424360
- [Background] Vanfleteren LEGW, Spruit MA, Wouters EFM, Franssen FME. Management of chronic obstructive pulmonary disease beyond the lungs. Lancet Respir Med. 2016 Nov;4(11):911-924. doi: 10.1016/S2213-2600(16)00097-7. Epub 2016 Jun 2. PMID 27264777
- [Background] Borel JC, Pepin JL, Pison C, Vesin A, Gonzalez-Bermejo J, Court-Fortune I, Timsit JF. Long-term adherence with non-invasive ventilation improves prognosis in obese COPD patients. Respirology. 2014 Aug;19(6):857-65. doi: 10.1111/resp.12327. Epub 2014 Jun 9. PMID 24912564
- [Background] Struik FM, Lacasse Y, Goldstein RS, Kerstjens HA, Wijkstra PJ. Nocturnal noninvasive positive pressure ventilation in stable COPD: a systematic review and individual patient data meta-analysis. Respir Med. 2014 Feb;108(2):329-37. doi: 10.1016/j.rmed.2013.10.007. Epub 2013 Oct 14. PMID 24157199